CLINICAL TRIAL: NCT06397352
Title: Effects of Buzzy® and ShotBlocker® on Pain, Anxiety and Satisfaction During the Administration of Tetanus-Diphtheria Vaccine to School-Aged Children: A Randomized Controlled Trial
Brief Title: Effects of Buzzy® and ShotBlocker® on Pain, Anxiety and Satisfaction During the Administration of Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hatice ERDEM ÖNDER, Research Assistant Dr., Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MehmetAkifU-SBF-HEÖ-02
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Pain; Anxiety; Satisfaction
Keywords: Buzzy; Shotblocker; pain; anxiety; satisfaction; vaccine
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to ShotBlocker®, Buzzy®, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShotBlocker® Group (Experimental): The ShotBlocker® is a small, flexible, drug-free plastic device with several short, blunt skin contact points on the bottom and a hole in the center through which injections can be administered. It is positioned onto the skin before an injection is made. After positioning the ShotBlocker® and ensuring that the contacts were in contact with the children's skin, the injection was made through the central hole by the nurse. The ShotBlocker® was cleaned with 70% alcohol before use on another child.
  Interventions: Other: ShotBlocker®
- Buzzy® Group (Experimental): Buzzy is a small plastic device powered by a vibrating motor and an ice pack. Buzzy is attached to the skin using a tourniquet 3 to 5 cm above the injection site just before the injection. Vibrations started 30 seconds before the procedure and continued until it was completed. The device was cleaned with 70% alcohol before use on another child.
  Interventions: Other: Buzzy® Group

INTERVENTIONS:
Other: ShotBlocker® — All children underwent a standard procedure. The standard procedure involved taking the child into the vaccination room, providing information about the vaccination procedure, introducing the researcher, and obtaining consent. The STAI-S was completed immediately before the vaccination. Children were assigned to groups as specified in the randomization procedure. The vaccination of children was performed by an experienced nurse working in the unit where the study was conducted to control for practitioner-related factors.It is positioned onto the skin before an injection is made. After positioning the ShotBlocker® and ensuring that the contacts were in contact with the children's skin, the injection was made through the central hole by the nurse. The ShotBlocker® was cleaned with 70% alcohol before use on another child.
  Arms: ShotBlocker® Group
Other: Buzzy® Group — All children underwent a standard procedure. The standard procedure involved taking the child into the vaccination room, providing information about the vaccination procedure, introducing the researcher, and obtaining consent. The STAI-S was completed immediately before the vaccination. Children were assigned to groups as specified in the randomization procedure. The vaccination of children was performed by an experienced nurse working in the unit where the study was conducted to control for practitioner-related factors. Vibrations started 30 seconds before the procedure and continued until it was completed. The device was cleaned with 70% alcohol before use on another child
  Arms: Buzzy® Group

SUMMARY:
The aim of this study was to detect and compare the effects of ShotBlocker® and Buzzy® methods on pain, anxiety, and satisfaction during the administration of Tetanus-Diphtheria vaccine to school-aged children. This study was an experimental randomized controlled trial. The sample was included 138 children in a family health centers aged 13 years who underwent Tetanus-Diphtheria vaccine. The participants were randomly assigned to ShotBlocker®, Buzzy®, and control groups. Each group included 46 children, of whom 23 were female and 23 were male. The State-Trait Anxiety Inventory and Visual Analog Scale were used to collect the data.

DETAILED DESCRIPTION:
This research aims to determine effects of Buzzy® and ShotBlocker® on pain and anxiety during the administration of tetanus-diphtheria vaccine to school-aged children.

The following hypotheses were determined for the present study. Hypothesis 1. ShotBlocker® is effective in reducing pain and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

Hypothesis 2. Buzzy® is effective in reducing pain and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

Hypothesis 3. Buzzy® is more effective than ShotBlocker in reducing pain and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

This prospective, randomised controlled study was conducted in one family health centers of Manisa, Turkey, between November 2021- August 2023. A parallel trial design was used describing, shotblocker, buzzy, and control group as the third arm. This study was guided by the Consolidated Standards of Reporting Trials (CONSORT) checklist. This study was conducted in one family health centers with the same nurse. Children aged 13 years who underwent tetanus- Diftevaccine injection were eligible to participate in the study. The inclusion criteria were being 13 years and being conscious (with the ability to communicate). The exclusion criteria were having a physical and psychological condition; taking any analgesics, sedatives, or anticonvulsants in the past 24 hours; having chronic or life-threatening disease; and refusing the shotblocker or buzzy intervention during vaccine injection. The sample size for the research was determined using G*power 3.0.8 software, and power analysis was conducted. With a 5% error rate, 80% power, and a medium effect size of 0.25 for the 3 groups with 2 repeated factors, it was calculated that 46 children should be taken for each group (Ellis, 2010). The study sample composed of 138 children. Childrens presenting for tetanus vaccine injection and fulfilling the inclusion criteria were assigned into three groups: Shotblocker®, Buzzy® and control groups (exposed to the conventional injection technique). So that effects of gender could be controlled, the childrens were first categorized according to their genders and then assigned into the three groups through block randomization. To ensure randomization and minimize all possible negative effects, the words shotblocker, buzzy and control, representing the three groups, were written on papers of the same color and shape and placed in a pink and a blue box. During the routine vaccination of children, which group would be included was determined by a lottery drawn by the child, just before the procedure started. The girls were asked to draw a paper from the pink box and boys from the blue box. This allowed keeping the effect of gender under control. Each group included 46 children, of whom 23 were female and 23 were male.

ELIGIBILITY:
Inclusion Criteria:

* 13 years
* being conscious (with the ability to communicate)

Exclusion Criteria:

* having a physical and psychological condition
* taking any analgesics, sedatives, or anticonvulsants in the past 24 hours
* having chronic or life-threatening disease
* refusing the shotblocker or buzzy intervention during vaccine injection.

Ages: 13 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Visual Analog Scale were completed immediately after the vaccination.
  This scale consists of a 10-cm line (0-10 cm or 0-100 mm). The 0-line on the scale indicates "no pain," and the 10-line indicates "unbearable pain." The child is asked to mark the place that expresses the degree of pain. The distance from the point marked by the child to the 0 line is measured to determine the degree of pain. In children aged 8 and above, the Visual Analog Scale (VAS) is considered the most reliable method.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | State-Trait Anxiety Inventory (STAI) were completed immediately after the vaccination
  The State-Trait Anxiety Inventory (STAI) has been employed in clinical settings to assess levels of both state (STAI-S; i.e., current) and trait (STAI-T; i.e., long-term, general) anxiety. This formwas developed by Spielberger et al. (1971) to measure the anxiety levels of children. The STAI-S was adapted into Turkish by Özusta in 1995, and its validity and reliability study was conducted. The inventory is a 3-point Likert-type scale consisting of 20 items that aim to evaluate feelings associated with state anxiety. The children evaluated how they felt 'at that moment' as "almost never" (1 point), "sometimes" (2 points), and "often" (3 points). The scale ranges from 20 to 60 points, with a high score indicating a high level of anxiety.
Satisfaction level | Satisfaction were completed immediately after the vaccination
  children were asked to rate their satisfaction level with the vaccination on a scale of 0 points "not satisfied" to 10 points "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Erdem Önder, Study Chair — Mehmet Akif Ersoy University; Dilek Sari, Study Director — Ege University; Nihal Taşkiran, Study Chair — Aydin Adnan Menderes University
Locations (1):
- Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No